CLINICAL TRIAL: NCT04524884
Title: The Efficacy and Safety of Anti-PD-1 Antibody Toripalimab Combined With Surufatinib for Locally Advanced Thyroid Cancer: a Phase II Study
Brief Title: Toripalimab Combined With Surufatinib for Locally Advanced Thyroid Cancer: a Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thca-NEO-ST
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Thyroid Cancer
Keywords: Toripalimab; Surufatinib; Thyroid cancer; Neoadjuvant therapy
MeSH Terms: conditions — Thyroid Neoplasms | interventions — surufatinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Surufatinib 250mg will be taken orally once daily continuously through a 21-day cycle of study treatment. Toripalimab 240mg will be intravenously administered on Day 1 of each cycle. After neoadjuvant Toripalimab and Surufatinib treatment, the patients will receive operation treatment if the tumor is evaluated as resectable cases by clinical examination.
  Interventions: Drug: Surufatinib; Drug: Toripalimab
- Cohort B (Experimental): Surufatinib 250mg will be taken orally once daily continuously through a 21-day cycle of study treatment. Toripalimab 240mg will be intravenously administered on Day 1 of each cycle. After neoadjuvant Toripalimab and Surufatinib treatment, the patients will receive further drug reatment, if the tumor is evaluated as unresectable cases and patients have potential benefits by clinical examination.
  Interventions: Drug: Surufatinib; Drug: Toripalimab
- Cohort C (Experimental): Surufatinib 250mg will be taken orally once daily continuously through a 21-day cycle of study treatment. Toripalimab 240mg will be intravenously administered on Day 1 of each cycle. After neoadjuvant Toripalimab and Surufatinib treatment, the patients will be removed from the study, if the tumor is evaluated as unresectable cases and patients have no potential benefits by clinical examination.
  Interventions: Drug: Surufatinib; Drug: Toripalimab

INTERVENTIONS:
Drug: Surufatinib — Surufatinib is a tablet in the form of 50mg, oral, once a day.
  Other Names: HMPL-012
Drug: Toripalimab — Toripalimab is an injection in the form of 240mg, intravenous, once three weeks.
  Other Names: JS001

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination of Toripalimab and Surufatinib for Locally Advanced Thyroid Cancer.

DETAILED DESCRIPTION:
Surufatinib (HMPL-012, previously named sulfatinib) is a small-molecule inhibitor targeting vascular endothelial growth factor receptors, fibroblast growth factor receptor 1 and colony-stimulating factor 1 receptor. A multi-center , opened, Phase II study have identified the efficacy and safety of Surufatinib in advanced medullary thyroid Carcinoma ( MTC) and iodine-refractory differentiated thyroid carcinoma (DTC).Toripalimab is a humanized immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed cell death 1 (programmed death-1; PD-1), with potential immune checkpoint inhibitory and antineoplastic activities. In the present study, we design a single-arm, single center Phase II trial to evaluate the efficacy and safety of the combination of Surufatinib wiht Toripalimab in locally advanced differentiated thyroid cancer as neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed an informed consent form and shows good compliance;
2. Age ≥18 years, male or female;
3. Pathologically diagnosed locally advanced differentiated thyroid cancer, including papillary thyroid cancer and follicular thyroid cancer;
4. Diagnosis of locally advanced disease should meet at least one of the criteria:1)Unresectable locally advanced lesion; 2)Difficult to achieve R0/R1 resection during preoperative assessment; 3)AJCC T4 stage: Primary tumor with invasion or adhesion of at least one of the following structures / organs, including: trachea, esophagus, common carotid artery, larynx, anterior vertebral fascia, brachial plexus;
5. Have at least one measurable lesion (RECIST 1.1);
6. Eastern Cooperative Oncology Group (ECOG) score 0-2;
7. Expected survival time ≥ 12 weeks;
8. If the patient presents with distant metastasis, the value of local treatment should be assessed by the investigator;
9. The patient volunteered to receive tumor biopsy/surgery during rull-in and rull-out periods.
10. The main organ functions meet the following criteria within 7 days before treatment:1)Standard blood test (without blood transfusion within 14 days):Hemoglobin (HB) ≥90g / L; Absolute neutrophil value (ANC) ≥ 1.5 × 109 / L; Platelet (PLT) ≥80 × 109 / L; 2)Biochemical inspection must meet the following standards: Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, if with liver metastases, ALT and AST ≤ 5 ULN; Serum creatinine (Cr) ≤ 1.5 ULN or creatinine clearance (CCr)>50ml / min; 3)International normalized ratio (INR) ≤2.3 or prothrombin time (PT) prolongs less than 6 seconds; 4)Urine routine indicates urinary protein <++, and the 24-hour urine protein quantification is less than 1.0 g.
11. Women of childbearing age should agree to use contraceptives during the study; negative serum or urine pregnancy tests within 14 days before study enrollment.

Exclusion Criteria:

1. History of a second malignancy during the past 5 years before inclusion in the study or during participation in the study, with the exception of a dermal basal cell or squamous cell carcinoma or cervical carcinoma in situ, if these were curatively treated;
2. Use any anti-tumor treatment within 4 weeks (28 days) prior to the start of the study treatment, except for TSH suppression treatment;
3. Previously used any immune checkpoint inhibitors, including but not limited to pembrolizumab, nivolumab, camrelizumab, sintilimab and etc;
4. With other uncontrolled cardiac symptoms or disease;
5. Patients whose blood pressure is still unsatisfactory with a blood pressure medication (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg) or a history of hypertensive encephalopathy or hypertensive crisis;
6. Those who have multiple factors (such as inability to swallow) that affect oral medication;
7. Patients with a gastrointestinal bleeding tendency including 1)Active peptic ulcer; 2)Fecal occult blood ≥ ++; 3)A history of hematemesis or melena within 3 months;
8. Coagulation disorder, such as INR greater than 1.5, or activated partial thromboplastin time (APTT) greater than 1.5 * ULN;
9. Significant hemoptysis within 2 months before screening, or the daily volume of hemoptysis reached half a teaspoon (2.5ml) or more;
10. Patients whose imaging showed that the tumor had invaded the important blood vessels or the researchers judged that the tumor was likely to invade important blood vessels during the subsequent study period and caused fatal bleeding;
11. Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism within 6 months;
12. Patients suffering from interstitial pneumonia or ILD, or with a history of interstitial pneumonia or ILD requiring hormone therapy, or with other pulmonary fibrosis，organic pneumonia(e.g., obliterative bronchiolitis), pneumoconiosis, drug-induced pneumonia and idiopathic pneumonia that may interfere with the diagnosis and management of immune-related pulmonary toxicity; or patients with CT image indicating active pneumonia or severely impaired pulmonary function during screening. Radiation pneumonia is acceptable in the radiation field. Patients with active tuberculosis will be excluded;
13. Active autoimmune disease or history of autoimmune disease with recurrence potential (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis): Patients with skin diseases that do not require systemic treatment such as vitiligo, psoriasis, hair loss, controlled type I diabetes receiving insulin therapy; childhood asthma that is completely relieved, or those who do not need any intervention in adulthood can be included; Patients with asthma who undergo medical intervention such as bronchiectasis, cannot be included;
14. Use immunosuppressive agents or systemic hormone therapy within preceding 14 days before the study starts to achieve the purpose of immunosuppression (dose>10mg/day prednisone or hormones with equivalent effects);
15. Patients who received strong CYP3A4/CYP2C19 inducer including rifampin (and its analogs) and hypericum perforatum or strong CYP3A4/CYP2C19 inhibitor within preceding 14 days;
16. Patients who have a history of severe allergies to any monoclonal antibody or anti-angiogenic targeted drugs;
17. Patients who have severe uncontrolled infection during study screening;
18. Patients who are pregnant or lactating;
19. Patients who refuse to receive tumor biopsy during rule-in and rule-out period;
20. Other reasons according to the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 16 months after the last patient enrolled
  Objective Response Rate

SECONDARY OUTCOMES:
R0/1 resection rate | Within one week after operation
  R0 and R1 resection rate reviewed by operation team and pathologists
DCR | 16 months after the last patient enrolled
  Disease Control Rate
TTR | 16 months after the last patient enrolled
  Time to objective response
PFS | 16 months after the last patient enrolled
  Progression Free Survival
OS | 16 months after the last patient enrolled
  Overall Survival
AE | From first dose to within 30 days after the last dose
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Qing-Hai Ji, MD, Principal Investigator — Fudan University; Yu-Long Wang, MD, Principal Investigator — Fudan University
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No